CLINICAL TRIAL: NCT04388397
Title: Immediate-access Arteriovenous Versus Standard Arteriovenous Grafts in Hemodialysis Patients: A Randomized Clinical Study
Brief Title: Immediate-access Arteriovenous Versus Standard Arteriovenous Grafts in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egyptian Biomedical Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 02090520
Record Dates: First submitted 2020-05-09; First posted 2020-05-14 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Hemodialysis Access Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate-access Arteriovenous Grafts (Experimental): Immediate-access Arteriovenous Grafts as a vascular access for hemodialysis patients
  Interventions: Procedure: Arteriovenous Grafts
- Standard Arteriovenous Grafts (Active Comparator): Standard Arteriovenous Grafts as a vascular access for hemodialysis patients
  Interventions: Procedure: Arteriovenous Grafts

INTERVENTIONS:
Procedure: Arteriovenous Grafts — Arteriovenous fistulae (AVF) are considered the main access for hemodialysis (HD). Arteriovenous grafts (AVGs) are an alternative access modality in patients with exhausted native venous access. Immediate-access arteriovenous grafts (IAAVGs) is a new modality in which dialysis can be started immediately to avoid complications of central venous catheters.

SUMMARY:
Arteriovenous fistulae (AVF) are considered the main access for hemodialysis (HD). Arteriovenous grafts (AVGs) are an alternative access modality in patients with exhausted native venous access. Immediate-access arteriovenous grafts (IAAVGs) is a new modality in which dialysis can be started immediately to avoid complications of central venous catheters.

DETAILED DESCRIPTION:
The study aimed to evaluate and compare patency rate and complications of standard arteriovenous grafts (SAVGs) and immediate-access arteriovenous grafts (IAAVGs) in end stage renal disease (ESRD) patients for one year after the intervention. Patients were randomly divided into two groups: SAVGs group and IAAVGs group. Patients with ESRD with no chance for native AVF were examined clinically and by duplex ultrasonography preoperatively. Follow up was for one year. Primary end points were the success rate, complications rate (hematoma, pseudo-aneurysm, graft site infection, systemic bacteremia), time of first cannulation. Secondary end points were primary and secondary patency within one year.

ELIGIBILITY:
Inclusion Criteria:

* Adult hemodialysis patients

Exclusion Criteria:

* Significant cardiorespiratory comorbidities.
* Peripheral vascular disease.
* Pregnancy or lactation.
* Severe bleeding disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 477 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Primary Patency | 1 year
  Patency of hemodialysis access
Success rate | 24 hours
  successful graft procedure

SECONDARY OUTCOMES:
Complications rate | 1 year
  Any graft complications

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Tawfik, PhD, Principal Investigator — Faculty of Medicine, Zagazig University
Locations (2):
- Egypt (2):
  - Faculty of Medicine, Zagazig University, Zagazig
  - Faculty of Medicine, Zagazig

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tawfik AM, Zidan MH, Salem A, Salem A. A randomized controlled study of early versus standard cannulation of arteriovenous grafts in hemodialysis patients. J Vasc Surg. 2022 Mar;75(3):1047-1053. doi: 10.1016/j.jvs.2021.08.106. Epub 2021 Sep 30. PMID 34601044